CLINICAL TRIAL: NCT03237676
Title: The Effect of Cognitive Rehabilitation Therapy in Improving Cognitive Function of Attention Following Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PO037-2015A
Record Dates: First submitted 2017-07-18; First posted 2017-08-02 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Mild Traumatic Brain Injury; Cognitive Impairment
Keywords: cognitive rehabilitation; diffusion tensor imaging; neuropsychology; functional outcome
MeSH Terms: conditions — Brain Concussion; Cognitive Dysfunction | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: intervention group receives structured cognitive rehabilitation therapy, control group receives conventional/pre-existing cognitive rehabilitation therapy.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are randomised on treatment arm. Co-investigators are blinded from knowing which participant receives which treatment arm.
  Cognitive outcome assessor is blinded from knowing which participant receives which treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualised structured cognitive rehabilitation therapy (Experimental): Participants of interventional arm will receive individualised structured cognitive rehabilitation therapy at the proposed health centre (University Malaya Medical Centre, Malaysia).
  Interventions: Other: Structured cognitive rehabilitation therapy
- Patient-centred cognitive therapy (Active Comparator): Participants of conventional arm will receive an existing cognitive rehabilitation treatment available at the proposed health centre (University Malaya Medical Centre, Malaysia).
  Interventions: Other: Patient-centred cognitive therapy

INTERVENTIONS:
Other: Structured cognitive rehabilitation therapy — A computer-based cognitive rehabilitation therapy Therapy frequency is one hour session per week for three months.
  Other Names: cognitive therapy; CogniPlus
  Arms: Individualised structured cognitive rehabilitation therapy
Other: Patient-centred cognitive therapy — Application of existing cognitive therapy at University Malaya Medical Centre, Malaysia. It is a patient-centred therapy approach over a period of three months, which include therapy session on symptoms management and coping strategies.
  Clinical and treatment review are provided as part of routine outpatient rehabilitation clinic review.
  Arms: Patient-centred cognitive therapy

SUMMARY:
This research is a randomised controlled study. The study hypothesis is cognitive rehabilitation for attention deficits following mild traumatic brain injury will improve patient's cognitive outcome, measured by neuropsychological and neuroimaging parameters. Participant recruitment is from University Malaya Medical Centre, Malaysia. All mild traumatic brain injury participants have to fulfil the study inclusion criteria and written consented for therapy. Control group receives existing patient-centred cognitive treatment whereas intervention group receives individualised structured cognitive rehabilitation therapy. The intervention begins at three months post injury and ends at six months post injury. Study outcome measurements are applied at pre and post treatment. This study was ethically approved by Medical Research Ethics Committee University Malaya Medical Centre (MREC ID NO: 2016928-4293).

DETAILED DESCRIPTION:
General study objective: to measure the effect of cognitive rehabilitation program for attention deficit applied in mild traumatic brain injury patients.

Specific objectives:

1. To measure the effect of a 12-week cognitive rehabilitation therapy for attention deficits in mild traumatic brain injury patients using neuropsychological and functional assessments.
2. To examine the correlation between neurocognitive deficits and structural brain changes at baseline and at six months post injury.

Study type and location: An interventional study conducted in University Malaya Medical Centre (UMMC), Malaysia.

Participants: Patients diagnosed with mild traumatic brain injury at Accident & Emergency Department in UMMC.

Outcome measures:

1. Neuropsychological Assessment Battery-Screening test
2. Diffusion Tensor Imaging parameters
3. Goal Attainment Scaling

Ethics approval: approved MREC ID NO: 2016928-4293

Consent: informed written consent will be obtained from all participants of research.

Estimated sample size:

Based on medium effect size Cohen's d = 0.35 Investigators used G*Power Version 3.1.9.2 for sample size calculation. Sample size calculated: 60 Estimating drop out rate of 40%=24. Therefore sample size target n= 84 mTBI patients.

Study design:

A two arm randomised controlled trial:

1. Mild traumatic brain injury control group, and
2. Mild traumatic brain injury intervention group.

The study protocol is divided into 3 segments:

1. Neurocognitive evaluation protocol:

   Investigators will perform Neuropsychological Assessment Battery-Screening test on both groups at three months and at six months following brain injury.
2. Imaging protocol:

   Investigators perform Diffusion Tensor Imaging for both groups at three months and at six months following brain injury.
3. Cognitive rehabilitation therapy protocol:

The focus is on attention deficits. Each study arm will receive different treatment approaches.

Mild traumatic brain injury control group will receive a patient-centred cognitive therapy. This is an application of existing cognitive rehabilitation treatment available at UMMC, which include therapy session on symptoms management and coping strategies. This is performed and monitored by a cognitive therapy trained Occupational Therapist. Clinical and treatment review are provided as part of routine outpatient rehabilitation clinic review.

Mild traumatic brain injury intervention group will receive individualised structured cognitive rehabilitation therapy that consist of:

1. Direct attention training:

   A deficit-oriented evidence-based treatment approach. The therapy for attention is computer-based and is divided into focused attention, selective attention, divided attention and sustained attention. Each treatment session is conducted by a trained Occupational Therapist in cognitive therapy and a rehabilitation medicine physician.
2. Strategic approach (metacognitive):

This involves generalisation of tasks to everyday functional skills. This approach is applied after each direct attention training session. This approach include review of individualised goals, review of cognitive related problem(s) encountered in participants daily activities since injury and problem-solving training. This is also performed by similar trained Occupational Therapist and reviewed by a rehabilitation medicine physician.

Randomisation sampling: Investigators apply simple randomisation in selection of mild traumatic brain injury control and intervention group participants.

ELIGIBILITY:
Inclusion Criteria:

* Mild traumatic brain injury as a result of motor vehicle accidents only.
* No previous history of head trauma.
* Education level of a minimum of 9 years (required for neuropsychological test).
* Normal Computed Tomography (CT) brain scan finding.
* Able to comply with cognitive rehabilitation therapy.
* No pre-existing chronic illness that can cause neurological complications, neurological diseases or psychiatric condition.
* Not on any regular medication that may alter or effect cognitive and psychological status.

Exclusion Criteria:

* Normal neuropsychological assessment test result at 3 months post injury (planned test time) for both study groups.
* Clinical evidence of alcohol influence at time of injury.
* Non Malaysian citizens
* Major polytrauma including long bone fractures, intra-abdominal injuries and chest injuries that require surgical and/or metal insertion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Neuropsychological Assessment Battery- Screening score | Perform at 3 months (pre-intervention) and 6 months (completed intervention) following mild traumatic brain injury
  Measure the change in score of Attention domain screening score and Total Screening Index Score at two different time points - 3 months and 6 months post brain injury.

SECONDARY OUTCOMES:
Change in Diffusion Tensor Imaging parameters | Perform at 3 months (pre-intervention) and 6 months (completed intervention) following mild traumatic brain injury
  Measure the change in mean values of white matter tract parameters at two different time points - 3 months and 6 months post brain injury.
Change in Goal Attainment Scaling score | Perform at 3 months (baseline) and 6 months (complete intervention) following mild traumatic brain injury
  Measure the change in Goal Attainment Scaling calculation score at two different time points - 3 months and 6 months post brain injury.

CONTACTS AND LOCATIONS:
Overall Officials: Norhamizan Hamzah, MBChB,MRehabMed, Principal Investigator — Rehabilitation Medicine Specialist, University of Malaya; Mazlina Mazlan, MBBS,MRehabMed, Study Chair — Consultant Rehabilitation Medicine & Associate Professor, University of Malaya; Vairavan Narayanan, MBBS,MSURG,FRCS, Study Chair — Consultant Neurosurgeon & Associate Professor, University of Malaya; Norlisah Ramli, MBBS,FRCR, Study Chair — Consultant Neuroradiologist & Professor, University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Veeramuthu V, Narayanan V, Kuo TL, Delano-Wood L, Chinna K, Bondi MW, Waran V, Ganesan D, Ramli N. Diffusion Tensor Imaging Parameters in Mild Traumatic Brain Injury and Its Correlation with Early Neuropsychological Impairment: A Longitudinal Study. J Neurotrauma. 2015 Oct 1;32(19):1497-509. doi: 10.1089/neu.2014.3750. Epub 2015 Jun 11. PMID 25952562
- [Background] Veeramuthu V, Narayanan V, Ramli N, Hernowo A, Waran V, Bondi MW, Delano-Wood L, Ganesan D. Neuropsychological Outcomes in Patients with Complicated Versus Uncomplicated Mild Traumatic Brain Injury: 6-Month Follow-Up. World Neurosurg. 2017 Jan;97:416-423. doi: 10.1016/j.wneu.2016.10.041. Epub 2016 Oct 15. PMID 27751922
- [Background] Veeramuthu V, Hariri F, Narayanan V, Tan LK, Ramli N, Ganesan D. Microstructural Change and Cognitive Alteration in Maxillofacial Trauma and Mild Traumatic Brain Injury: A Diffusion Tensor Imaging Study. J Oral Maxillofac Surg. 2016 Jun;74(6):1197.e1-1197.e10. doi: 10.1016/j.joms.2016.01.042. Epub 2016 Jan 30. PMID 26917201
- [Background] Marshall S, Bayley M, McCullagh S, Velikonja D, Berrigan L, Ouchterlony D, Weegar K; mTBI Expert Consensus Group. Updated clinical practice guidelines for concussion/mild traumatic brain injury and persistent symptoms. Brain Inj. 2015;29(6):688-700. doi: 10.3109/02699052.2015.1004755. Epub 2015 Apr 14. PMID 25871303
- [Background] Carroll LJ, Cassidy JD, Cancelliere C, Cote P, Hincapie CA, Kristman VL, Holm LW, Borg J, Nygren-de Boussard C, Hartvigsen J. Systematic review of the prognosis after mild traumatic brain injury in adults: cognitive, psychiatric, and mortality outcomes: results of the International Collaboration on Mild Traumatic Brain Injury Prognosis. Arch Phys Med Rehabil. 2014 Mar;95(3 Suppl):S152-73. doi: 10.1016/j.apmr.2013.08.300. PMID 24581903
- [Background] Cassidy JD, Cancelliere C, Carroll LJ, Cote P, Hincapie CA, Holm LW, Hartvigsen J, Donovan J, Nygren-de Boussard C, Kristman VL, Borg J. Systematic review of self-reported prognosis in adults after mild traumatic brain injury: results of the International Collaboration on Mild Traumatic Brain Injury Prognosis. Arch Phys Med Rehabil. 2014 Mar;95(3 Suppl):S132-51. doi: 10.1016/j.apmr.2013.08.299. PMID 24581902
- [Background] Hulkower MB, Poliak DB, Rosenbaum SB, Zimmerman ME, Lipton ML. A decade of DTI in traumatic brain injury: 10 years and 100 articles later. AJNR Am J Neuroradiol. 2013 Nov-Dec;34(11):2064-74. doi: 10.3174/ajnr.A3395. Epub 2013 Jan 10. PMID 23306011
- [Background] das Nair R, Lincoln NB, Ftizsimmons D, Brain N, Montgomery A, Bradshaw L, Drummond A, Sackley C, Newby G, Thornton J, Stapleton S, Pink A. Rehabilitation of memory following brain injury (ReMemBrIn): study protocol for a randomised controlled trial. Trials. 2015 Jan 6;16:6. doi: 10.1186/1745-6215-16-6. PMID 25559090
- [Background] Temple RO, Zgaljardic DJ, Abreu BC, Seale GS, Ostir GV, Ottenbacher KJ. Ecological validity of the neuropsychological assessment battery screening module in post-acute brain injury rehabilitation. Brain Inj. 2009 Jan;23(1):45-50. doi: 10.1080/02699050802590361. PMID 19096970
- [Background] Zgaljardic DJ, Temple RO. Reliability and validity of the Neuropsychological Assessment Battery-Screening Module (NAB-SM) in a sample of patients with moderate-to-severe acquired brain injury. Appl Neuropsychol. 2010 Jan;17(1):27-36. doi: 10.1080/09084280903297909. PMID 20146119
- [Derived] Hamzah N, Narayanan V, Ramli N, Mustapha NA, Mohammad Tahir NA, Tan LK, Danaee M, Muhamad NA, Drummond A, das Nair R, Goh SY, Mazlan M. Randomised controlled clinical trial of a structured cognitive rehabilitation in patients with attention deficit following mild traumatic brain injury: study protocol. BMJ Open. 2019 Sep 18;9(9):e028711. doi: 10.1136/bmjopen-2018-028711. PMID 31537559